CLINICAL TRIAL: NCT00872729
Title: A Pilot Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Cysteamine Bitartrate Delayed-release Capsules (RP103), Compared to Cysteamine Bitartrate (Cystagon®) in Patients With Nephropathic Cystinosis
Brief Title: Pilot Study of Safety, Tolerability, Pharmacokinetics/Pharmacodynamics of RP103 Compared to Cystagon® in Patients With Cystinosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-01
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Cystinosis
Keywords: cystinosis; cysteamine; inheritable disease; orphan disease; CTNS protein, human; nephropathic cystinosis
MeSH Terms: conditions — Cystinosis; Rare Diseases | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystagon® (Active Comparator): Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules, 150 mg/50 mg
  Interventions: Drug: Cystagon®
- RP103 (Experimental): Test Product: RP103 (Cysteamine Bitartrate) Delayed-release Capsules, 75 mg
  Interventions: Drug: RP103

INTERVENTIONS:
Drug: Cystagon® — Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules, 150 mg/50 mg.
  Duration of Treatment and Dose: Reference Period up to four doses Q6H.
  Arms: Cystagon®
Drug: RP103 — Test Product: RP103 (Cysteamine Bitartrate) Delayed-release Capsules, 75 mg.
  Duration of treatment and Dose: Single dose of Test Product at dose equivalent to Reference Product.
  Arms: RP103

SUMMARY:
Cystinosis is an inheritable disease that if untreated, results in kidney failure as early as the first decade of life. The current marketed therapy is Cystagon® (cysteamine bitartrate) which must be taken every six hours for the rest of the patient's life to prevent complications of cystinosis. RP103 is a formulation of cysteamine bitartrate that is being studied to see if it may be able to be given less frequently, once every 12 hours, and have similar results.

DETAILED DESCRIPTION:
This is a single-dose, open-labeled, non-randomized, two-period study of Cysteamine Bitartrate Delayed-release Capsules (RP103) and Cystagon® in up to 10 patients (male or female) with nephropathic cystinosis under fasting conditions. It will involve a 4 night check-in to a clinical research center.

Study with completed results acquired from Horizon in 2024

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must have nephropathic cystinosis.
* Children less than 22.5 kg will only be included in the study if the investigator feels they can safely participate in the study including the required blood draw volume for the safety and PK/PD assessments.
* Subjects must be on a stable dose of Cystagon® at least 21 days prior to Screening.
* Subjects must be able to swallow a 150 mg Cystagon® capsule with the capsule intact.
* Within the last 2 months, no clinically significant change in liver function [i.e., ALT, AST, alkaline phosphatase, bilirubin (total and direct)] and renal function [i.e., serum creatinine, albumin, total protein] at Screening as determined by the Investigator.
* Sexually active female subjects of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy] or at least 2 years naturally postmenopausal) must agree to utilize the same acceptable form of contraception from screening through completion of the study.
* Subjects or their authorized caregiver must provide written informed consent and assent (where applicable) prior to participation in the study.
* If in the opinion of the investigator, patients can safely provide the study required blood draw volume.
* Subjects must be willing and able to comply with the study restrictions and requirements.

Exclusion Criteria:

* If, in the opinion of the investigator, the planned study dose would exceed the patient's tolerability of cysteamine based on their prior Cystagon® steady state drug requirements.
* Evidence of or verbal attestation of Helicobacter pylori infection, presently, or within the last 90 days prior to Screening.
* Subjects with a known history, currently or within the past 90 days prior to Screening, of the following conditions or other health issues that make it, in the opinion of the investigator, unsafe for them to participate, or whose concomitant medical problems preclude them from committing to the study schedule including the following: Crohn's disease, inflammatory bowel disease (if currently active) or have had prior resection of small intestine; • History of heart disease, e.g., myocardial infarction, heart failure, arrhythmias; Any bleeding disorder; Malignant disease; Severe liver disease as defined as ALT or AST > 2 times the upper limit of normal.
* Subjects who have had a kidney transplant.
* Subjects who are planning or are a registered candidate for a kidney transplant within 3 months of the Screening or have a serum creatinine > 2.4.
* Subjects with known hypersensitivity to cysteamine.
* If female (of child-bearing potential), are nursing, planning a pregnancy, known or suspected to be pregnant, or have a positive urine pregnancy screen.
* Patients with a hemoglobin level < 10.5.
* Subjects who have a made a blood donation within 60 days prior to study initiation.
* Subjects who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- University of California San Diego Medical Center, San Diego, California, United States

REFERENCES:
- [Background] Dohil R, Fidler M, Barshop BA, Gangoiti J, Deutsch R, Martin M, Schneider JA. Understanding intestinal cysteamine bitartrate absorption. J Pediatr. 2006 Jun;148(6):764-9. doi: 10.1016/j.jpeds.2006.01.050. PMID 16769383
- [Background] Fidler MC, Barshop BA, Gangoiti JA, Deutsch R, Martin M, Schneider JA, Dohil R. Pharmacokinetics of cysteamine bitartrate following gastrointestinal infusion. Br J Clin Pharmacol. 2007 Jan;63(1):36-40. doi: 10.1111/j.1365-2125.2006.02734.x. PMID 17229040
- [Background] Levtchenko EN, van Dael CM, de Graaf-Hess AC, Wilmer MJ, van den Heuvel LP, Monnens LA, Blom HJ. Strict cysteamine dose regimen is required to prevent nocturnal cystine accumulation in cystinosis. Pediatr Nephrol. 2006 Jan;21(1):110-3. doi: 10.1007/s00467-005-2052-0. Epub 2005 Oct 27. PMID 16252107
- See also: RP103 (marketed as PROCYSBI) is now approved by the US FDA for management of nephropathic cystinosis in patients 6 years and older — http://www.procysbi.com
- See also: Click here for more information about UCSD's cystinosis program — http://biochemgen.ucsd.edu/Cystinosis/Index.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystagon® and RP103: Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules,150 mg/50 mg; Test Product: RP103 (Cysteamine Bitartrate) Delayed-release Capsules,75 mg; Single-dose, open-label, nonrandomized, 2-period, crossover study of cysteamine bitartrate delayed-release capsules (RP103) and Cystagon®. Subjects were enrolled sequentially and received Cystagon® first followed by RP103.
Period: Overall Study
Arm/Group | Cystagon® and RP103
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cystagon® and RP103: Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules,150 mg/50 mg; Test Product: RP103 (Cysteamine Bitartrate) Delayed-release Capsules,75 mg.
Arm/Group | Cystagon® and RP103
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pharmacokinetic Parameter: Cmax of Cysteamine
Time Frame: 12 hours post RP103 dosing and 7 hours post 1st Cystagon® dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 9 | 9
umol/L | 42.02 (51) | 33.06 (55)

2. Primary Outcome: Plasma Pharmacokinetic Parameter: Tmax of Cysteamine
Time Frame: 12 hours post RP103 dosing and 7 hours post 1st Cystagon® dosing
Measure: Median (Full Range); unit: hour
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 9 | 9
hour | 1.00 [0.50 to 2.00] | 3.00 [0.00 to 5.13]

3. Primary Outcome: Plasma Pharmacokinetic Parameter: AUC(0-t) of Cysteamine
Description: t = 6 for Cystagon and t = 12 for RP103. Cystagon is dosed every 6 hours and there is no measurement after 6 hours and up to 12 hours.
Time Frame: 12 hours post RP103 dosing and 6 hours post 1st Cystagon® dosing
Population: Subjects were enrolled sequentially according to the study design. A mixed-effects linear model was used to assess differences between the RP103 and Cystagon treatment groups. Sample size is based on feasibility rather than statistical considerations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol•h/L
Arm/Group | Cystagon® | RP103
Number analyzed (Participants) | 9 | 9
umol•h/L | 107.89 (58) | 119.17 (46)

4. Primary Outcome: Pharmacodynamic Parameter: Changes of White Blood Cell (WBC) Cystine Level From Baseline
Description: The pharmacodynamic (PD) parameter measures the changes of WBC cystine level from the baseline.
  Cystine is a disulfide amino acid formed through oxidation of two molecules of cysteine; hence, cystine's concentration is commonly given in half-cystine equivalents to avoid confusion.
  The level of cystine in WBC/leukocytes is expressed in units of nmol half-cystine/mg protein (nmol ½ cystine/mg protein). Half-cystine is quantified by a reduction of cystine followed by an assay for cysteine, which is then normalized by the total cellular protein content within the sample using methods of such as Lowry assay, bicinchoninic acid assay, or Bradford.
Time Frame: up to 12 hours post Cystagon® dosing and RP103 dosing
Population: Sample size is based on feasibility rather than statistical considerations. Analysis time differences (0-6 hours) is due to different absorption characteristics of Cysteamine between RP103 and Cystagon. Cystagon is dosed every 6 hours and there is no measurement after 6 hours and up to 12 hours.
Measure: Mean (Standard Deviation); unit: nmol 1/2 cystine/mg protein
Groups:
- Cystagon® (0.5 Hour); Cystagon® (1 Hour); Cystagon® (2 Hour); Cystagon® (2.5 Hour); Cystagon® (3 Hour); Cystagon® (4 Hour); Cystagon® (6 Hour); Cystagon® (8 Hour); Cystagon® (10 Hour); Cystagon® (12 Hour): Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules, 150 mg/50 mg.
- RP103 (0.5 Hour); RP103 (1 Hour); RP103 (2 Hour); RP103 (2.5 Hour); RP103 (3 Hour); RP103 (4 Hour); RP103 (6 Hour); RP103 (8 Hour); RP103 (10 Hour); RP103 (12 Hour): Test Product: RP103 (Cysteamine Bitartrate) Delayed-release Capsules, 75 mg.
Arm/Group | Cystagon® (0.5 Hour) | RP103 (0.5 Hour) | Cystagon® (1 Hour) | RP103 (1 Hour) | Cystagon® (2 Hour) | RP103 (2 Hour) | Cystagon® (2.5 Hour) | RP103 (2.5 Hour) | Cystagon® (3 Hour) | RP103 (3 Hour) | Cystagon® (4 Hour) | RP103 (4 Hour) | Cystagon® (6 Hour) | RP103 (6 Hour) | Cystagon® (8 Hour) | RP103 (8 Hour) | Cystagon® (10 Hour) | RP103 (10 Hour) | Cystagon® (12 Hour) | RP103 (12 Hour)
Number analyzed (Participants) | 6 | 0 | 3 | 3 | 6 | 0 | 0 | 6 | 3 | 3 | 6 | 6 | 9 | 6 | 0 | 3 | 0 | 3 | 3 | 6
nmol 1/2 cystine/mg protein | 0.11 (0.24) |  | -0.10 (0.02) | 0.87 (0.33) | -0.07 (0.28) |  |  | 0.19 (0.48) | -0.14 (0.06) | 0.43 (0.70) | -0.01 (0.15) | 0.10 (0.50) | 0.30 (0.34) | 0.22 (0.41) |  | 0.20 (0.31) |  | 0.45 (0.36) | 0.37 (0.18) | 0.72 (0.47)

ADVERSE EVENTS:
Time Frame: After a dose of study drug (RP103 or Cystagon®) on or after study entry, for up to 10 days.
Groups:
- Cystagon®: Reference Product: Cystagon® (Cysteamine Bitartrate) Capsules, 150 mg/50 mg;
Arm/Group | Cystagon® | RP103
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/9 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cystagon® (N=9) | RP103 (N=9)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breath odor (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 3 (4) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may publish or disclose study data, with the restriction that sponsor may embargo such communications for a period up to 60 days from the time submitted to sponsor.